CLINICAL TRIAL: NCT05724069
Title: Velusetrag for the Treatment of Chronic Intestinal Pseudo-Obstruction (CIPO). A Multicenter, Double-blind, Placebo-controlled, Cross-over, Multiple (n=1) Trial.
Brief Title: Velusetrag for the Treatment of Chronic Intestinal Pseudo-Obstruction (CIPO).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VE-CIP2001/2021
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Intestinal Pseudo-obstruction
MeSH Terms: interventions — TD-5108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence A (Other): Eligible subjects will be treated for 4 periods with either velusetrag 15 mg once a day (2 periods) or placebo (2 periods), with a wash-out period of 2 weeks between treatment periods.
  The progression order of this sequence is: velusetrag first intervention 4 weeks, 2 weeks of wash-out period, then second intervention of placebo for 4 weeks, 2 weeks of wash-out period, then third intervention of velusetrag for other 4 weeks, 2 weeks of wash-out period and last 4 weeks of placebo as fourth intervention.
  Interventions: Drug: Velusetrag 15 mg once daily for 4 weeks.; Drug: Placebo once daily for 4 weeks.
- Sequence B (Other): Eligible subjects will be treated for 4 periods with either velusetrag 15 mg once a day (2 periods) or placebo (2 periods), with a wash-out period of 2 weeks between treatment periods.
  The progression order of this sequence is: placebo first intervention 4 weeks, 2 weeks of wash-out period, then second intervention of velusetrag for 4 weeks, 2 weeks of wash-out period, then third intervention of placebo for other 4 weeks, 2 weeks of wash-out period and last 4 weeks of velusetrag as fourth intervention.
  Interventions: Drug: Velusetrag 15 mg once daily for 4 weeks.; Drug: Placebo once daily for 4 weeks.
- Sequence C (Other): Eligible subjects will be treated for 4 periods with either velusetrag 15 mg once a day (2 periods) or placebo (2 periods), with a wash-out period of 2 weeks between treatment periods.
  The progression order of this sequence is: velusetrag first intervention 4 weeks, 2 weeks of wash-out period, then second intervention of placebo for 4 weeks, 2 weeks of wash-out period, then third intervention of placebo for other 4 weeks, 2 weeks of wash-out period and last 4 weeks of velusetrag as fourth intervention.
  Interventions: Drug: Velusetrag 15 mg once daily for 4 weeks.; Drug: Placebo once daily for 4 weeks.
- Sequence D (Other): Eligible subjects will be treated for 4 periods with either velusetrag 15 mg once a day (2 periods) or placebo (2 periods), with a wash-out period of 2 weeks between treatment periods.
  The progression order of this sequence is: placebo first intervention 4 weeks, 2 weeks of wash-out period, then second intervention of velusetrag for 4 weeks, 2 weeks of wash-out period, then third intervention of velusetrag for other 4 weeks, 2 weeks of wash-out period and last 4 weeks of placebo as fourth intervention.
  Interventions: Drug: Velusetrag 15 mg once daily for 4 weeks.; Drug: Placebo once daily for 4 weeks.

INTERVENTIONS:
Drug: Velusetrag 15 mg once daily for 4 weeks. — Subjects will be randomly allocated in a blinded fashion to 1 out of the 4 treatment sequences (each sequence include 4 periods, 2 periods with velusetrag and 2 periods with placebo). There will be a wash-out period between each treatment period.
Drug: Placebo once daily for 4 weeks. — Subjects will be randomly allocated in a blinded fashion to 1 out of the 4 treatment sequences (each sequence include 4 periods, 2 periods with velusetrag and 2 periods with placebo). There will be a wash-out period between each treatment period.

SUMMARY:
This is a phase II, multicenter, double-blind, placebo-controlled trial to evaluate the efficacy and safety of velusetrag once a day, compared to placebo, in subjects with CIPO.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with history of chronic idiopathic intestinal pseudo-obstruction or CIPO secondary to neurodegenerative or demyelinating disease.
* Subjects with estimated oral caloric intake of at least 30% of the daily age- and sex-recommended caloric intake.
* Subjects with at least 2 out of 4 CIPO gastrointestinal symptoms each of the 2 with a score ≥3 (on a 0 to 4 scale) at Day -1
* Subjects accepting to provide and legally capable of providing free and informed consent to all procedures included in the protocol.
* All sexually active male participants who are partner of women of childbearing potential must use condom during intercourse until the 90th day after the end of the entire study.
* Female participants are eligible if they are: i) of non-childbearing potential or ii) of childbearing potential with a negative pregnancy test result at screening and randomization AND agreeing to use a highly effective method of contraception (i.e., with failure rate of less than 1% per year) until the end of the entire study.

Exclusion Criteria:

* Subjects with primary CIPO or CIPO secondary to other known endocrine/metabolic, autoimmune diseases and neurologic conditions other than neurodegenerative or demyelinating diseases.
* Subjects with conditions characterized by mechanical intestinal obstruction.
* Nasogastric tube, gastrostomy tube, or jejunostomy feeding tube in place at randomization or planned throughout the duration of the study, or artificial food need scale stage 3.
* Presence of untreated clinically relevant thyroid dysfunction or known thyroid dysfunction not well controlled by treatment deemed clinically significant by the Investigator.
* Subjects with history of diabetes at screening.
* Clinically significant ECG abnormalities at screening and randomization.
* Screening ECG with a QTcF >450 msec in males or >470 msec in females or family history of sudden cardiac death.
* Subjects requiring a low galactose diet.
* Hypersensitivity or documented intolerance to lactulose, lactose or any excipient of the lactulose preparation to be used for L-BT.
* History of sensitivity to velusetrag, or any of the velusetrag or placebo excipients.
* Use of scopolamine or erythromycin within 2 weeks prior to screening and/or planned throughout the duration of the study.
* Use of 5-HT4 receptor agonists within 5 days prior to randomization and/or planned throughout the duration of the study
* Use of opioids within 8 weeks from screening and/or planned throughout the duration of the study.
* Received strong cytochrome P450-isozyme 3A4 (CYP3A4) inhibitors within 2 weeks prior to screening and/or planned throughout the duration of the study.
* Received strong P-glycoprotein (P-gp) transporter inhibitors within 2 weeks prior to Screening and/or planned throughout the duration of the study.
* Received strong breast cancer resistance protein transporter inhibitors within 2 weeks prior to screening and/or planned throughout the duration of the study.
* Current swab-positive or suspected (under investigation) COVID-19 infection.
* Cancer (excluding non-melanoma skin cancer) and/or need of any anti-cancer treatment (also including radiotherapy) within the last 5 years.
* Severe kidney impairment.
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) levels >2.5 times the upper limit of normal (ULN); bilirubin (unless deemed to be due to Gilbert's Syndrome) or alkaline phosphatase (ALP) >1.5 times ULN.
* Severe hepatic impairment defined as Child-Pugh C.
* History of any of the following cardiac disorders: i) torsade de pointes, ventricular tachycardia, ventricular fibrillation; ii) previous myocardial infarction, unstable angina pectoris, acute coronary syndrome, coronary artery or cerebral revascularization procedure or stroke within the previous 18 months; iii) angina pectoris class 2-4 during the last 12 months prior to screening; iv) congestive heart failure NYHA class III-IV during the last 18 months prior to screening.
* History of any alcohol or drug abuse or dependence within the last year (Investigator's judgement).
* Any current significant health condition that in the Investigator's judgement may: i) jeopardize the patient's safe participation in the trial or ii) make unlikely the patient's completion of the study or iii) make unlikely the patient's compliance with the study procedures.
* Pregnant or breastfeeding woman.
* Use of any experimental drug within 12 weeks prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven Gasthuisberg Campus, Leuven, Belgium
- Italy (2):
  - Policlinico S.Orsola-Malpighi, Bologna
  - Aou Arcispedale Sant'Anna Di Cona, Cona
- Hospital General Vall Hebron, Barcelona, Spain

REFERENCES:
- [Derived] Malagelada C, De Giorgio R, Cogliandro RF, Alcala-Gonzalez L, Costanzini A, Scuderi V, Manzoni S, Pasquali E, Tack J, Stanghellini V. Clinical Trial: Efficacy and Safety of Velusetrag in Chronic Intestinal Pseudo-Obstruction: A Randomized, Phase 2, Placebo-Controlled, Crossover, Multiple (n = 1), Proof-of-Concept Study. Neurogastroenterol Motil. 2026 Jan;38(1):e70246. doi: 10.1111/nmo.70246. PMID 41553253

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A; Sequence B; Sequence C; Sequence D: Eligible subjects will be treated for 4 periods with either velusetrag (2 periods) or placebo (2 periods), with a wash-out period of 2 weeks between treatment periods.
  The progression order of the treatment periods varies in each sequence.
  Velusetrag: Subjects will be randomly allocated in a blinded fashion to 1 out of the 4 treatment sequences (each sequence include 4 periods, 2 periods with velusetrag and 2 periods with placebo). There will be a wash-out period between each treatment period.
  Placebo: Subjects will be randomly allocated in a blinded fashion to 1 out of the 4 treatment sequences (each sequence include 4 periods, 2 periods with velusetrag and 2 periods with placebo). There will be a wash-out period between each treatment period.
Period: Overall Study
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D
Started | 5 (5 subjects started the first intervention period in sequence A) | 4 (4 subjects started the first intervention period in sequence B) | 4 (4 subjects started the first intervention period in sequence C) | 4 (4 subjects started the first intervention period in sequence D)
Completed | 5 (5 subjects completed the fourth intervention period in sequence A) | 4 (4 subjects completed the fourth intervention perion in sequence B) | 4 (4 subjects completed the fourth intervention period in sequence C) | 3 (3 subjects completed the fourth intervention period in sequence D as 1 withdrawal after the first intervention period)
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: demographic characteristics are summarized descriptively overall
Arm/Group | Overall
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 11
  Spain | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Weekly Global Gastrointestinal Symptoms Average Index Score (WGGSAIS).
Description: Mean change in weekly global gastrointestinal symptoms average index score (WGGSAIS) from pretreatment (PRE) to the end of each treatment period (EOT). The weekly global gastrointestinal symptoms average index score is obtained by averaging the scores for each of the 4 symptoms, abdominal pain, bloating, nausea and vomiting, assessed using a subject's e-diary. Each symptom was rated using a recall period of 7 days and a Likert scale with the following categories: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe according to its influence on usual activity. The WGGSAIS thus ranges between 0 and 4 with lower scores representing better health.
Time Frame: 4 weeks. The change is derived as the end of treatment period minus the pre-treatment value of the period, for each period.
Population: Modified Full Analysis Set 1 (mFAS1): the set of subjects responder/naïve to 5-HT4 agonist randomized and treated who reported data on the primary endpoint at least once during a velusetrag treatment period and at least once during a placebo treatment period. Arms were not mutually exclusive.
Measure: Mean (Standard Deviation); unit: score
Groups:
- Modified Full Analysis Set 1 Velusetrag: The velusetrag arm includes all subjects who took velusetrag during the 4 periods/4 sequences crossover, multiple (n=1) trial.
- Modified Full Analysis Set 1 Placebo: The Placebo arm includes all subjects who took placebo during the 4 periods/4 sequences cross-over, multiple (n=1) trial.
Arm/Group | Modified Full Analysis Set 1 Velusetrag | Modified Full Analysis Set 1 Placebo
Number analyzed (Participants) | 15 | 15
score | -0.424 (0.6926) | -0.185 (0.6876)
Statistical Analysis 1: Comparison: Modified Full Analysis Set 1 Velusetrag vs Modified Full Analysis Set 1 Placebo; Subjects in this analysis are 15 and not 30 (this happens because arms are not mutually exclusive, as explained in previous sections). Each subject can contribute with 0, 1, 2 pairs. Only data that constitute pairs evaluable for primary endpoint are considered in the analysis; the pairs evaluable for primary endpoint were 23; Test type: Superiority; p = 0.1279, paired T-test; Median Difference (Net) = -0.239, 95% CI 2-sided [-0.553 to 0.074]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Velusetrag 15 mg Once a Day | Placebo Once a Day
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 7/17 | 10/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velusetrag 15 mg Once a Day (N=17) | Placebo Once a Day (N=17)
hypertension (Vascular disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Anemia Vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (2) | 1 (1)
Eye swelling (Eye disorders) | 1 (2) | 1 (5)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contracturer (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT05724069/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT05724069/SAP_001.pdf